CLINICAL TRIAL: NCT05574400
Title: The Caffeine, Postoperative Delirium, and Change in Outcomes After Surgery (CAPACHINOS-2) Study
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University of Michigan (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Principal Investigator, Phillip Vlisides, Assistant Professor of Anesthesiology, University of Michigan
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: HUM00218290; R01AG075005 (NIH)
Record Dates: First submitted 2022-10-06; First posted 2022-10-10 (Actual); Last update posted 2025-07-24 (Actual); Status verified 2025-07

CONDITIONS: Postoperative Delirium; Postoperative Cognitive Dysfunction; Mild Cognitive Impairment
Keywords: Postoperative Delirium; Neurocognitive Disorders; Mild Cognitive Impairment; Alzheimer's Disease
MeSH Terms: conditions — Emergence Delirium; Postoperative Cognitive Complications; Cognitive Dysfunction; Neurocognitive Disorders; Alzheimer Disease | interventions — caffeine citrate

STUDY DESIGN:
Intervention Model Description: This will be a three-arm parallel trial.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: This will be a single-center, quadruple-blinded, randomized control trial at Michigan Medicine
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- Control (Placebo Comparator): Prepared intravenous piggyback solution of 5 percent dextrose water at multiple postoperative time points over a 30-minute infusion period.
  Interventions: Drug: Dextrose Water
- Low-dose Caffeine (Experimental): Prepared intravenous low-dose caffeine citrate (1.5 mg/kg) at multiple postoperative time points over a 30-minute infusion period.
  Interventions: Drug: Caffeine citrate
- High-dose Caffeine (Experimental): Prepared intravenous high-dose caffeine citrate (3 mg/kg) at multiple postoperative time points over a 30-minute infusion period.
  Interventions: Drug: Caffeine citrate

INTERVENTIONS:
Drug: Dextrose Water — Dextrose 5% in water
  Arms: Control
Drug: Caffeine citrate — Low-dose caffeine citrate (1.5 mg/kg)
  Arms: Low-dose Caffeine
Drug: Caffeine citrate — High-dose Caffeine citrate (3 mg/kg)
  Arms: High-dose Caffeine

SUMMARY:
The objective of this study is to test the effects of caffeine on neurocognitive and clinical recovery after major surgery. Specifically, this trial tests the primary hypothesis that caffeine will reduce the incidence of postoperative delirium.

DETAILED DESCRIPTION:
Delirium is a syndrome characterized by failure of basic cognitive functions that affects approximately 20-50% of older surgical patients. Delirium during surgical recovery is associated with increased mortality, cognitive and functional decline, and prolonged hospitalization. In fact, 3-year survival rates for acutely hospitalized patients with delirium, and subsyndromal delirium, are both less than 50%. Older age is predictive of delirium after surgery, and with aging surgical populations, the incidence of postoperative delirium and related complications are likely to increase in the coming years.

Caffeine represents a novel, neurobiologically informed candidate intervention for reducing risk of early postoperative delirium. Caffeine promotes arousal via adenosine receptor antagonism and improves cognitive function concurrent with increased cortical cholinergic tone. Our preliminary data suggest that caffeine reduces risk of postanesthesia care unit (PACU) delirium in adult non-cardiac surgery patients by optimizing cortical dynamics for cognition. Caffeine also optimizes key neurocognitive processes that support information processing and may improve other, related aspects of clinical recovery, such as rebound headache in habitual caffeine users. The objective of this trial is to thus test the effects of caffeine on neurocognitive and clinical recovery after major surgery. Specifically, the primary hypothesis is that caffeine will reduce the incidence of postoperative delirium. The secondary objectives are to (1) test whether caffeine positively impacts the quality of postoperative recovery via validated patient-reported measures and (2) identify neural correlates of delirium and Mild Cognitive Impairment via advanced electroencephalographic (EEG) analysis.

ELIGIBILITY:
Inclusion Criteria:

1. Adult (>/= 70 years old) undergoing non-cardiac, non-intracranial neurologic, non-major vascular surgery requiring general anesthesia with a planned admission for at least 48 hours.
2. Stated willingness to comply with all study procedures and availability for the duration of the study.
3. Provision of signed and dated informed consent form.

Exclusion Criteria:

1. Emergency surgery
2. Outpatient surgery
3. Severe cognitive impairment precluding the capacity for informed consent
4. Seizure disorder history
5. Intolerance or allergy to caffeine (based on subjective reporting or objective documentation)
6. Weight >130 kg (as a 3 mg/kg dose would approach the upper limit of daily intake recommended by the FDA)
7. Enrollment in conflicting research study
8. Patients in acute liver failure
9. Acute kidney injury preoperatively
10. Diagnosis of pheochromocytoma
11. Active carcinoid syndrome
12. Severe audiovisual impairment
13. Non-English speaking

Min Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 250 (Estimated)
Dates: Start 2023-02-20 (Actual); Primary Completion 2026-04-30 (Estimated); Study Completion 2026-05-31 (Estimated)

PRIMARY OUTCOMES:
Delirium | Day of surgery through afternoon of postoperative day three
  Any positive delirium screen (yes/no) as determined by the long-form Confusion Assessment Method (CAM), and supplemented by a validated daily chart review method.

SECONDARY OUTCOMES:
Delirium Severity | Day of surgery through afternoon of postoperative day three
  For all participants screened for delirium, the associated severity score will be recorded using the Confusion Assessment Method Long Form Severity Score (CAM-S) (n, 0-19, with higher number indicating more severe delirium)
Delirium Duration | Day of surgery through afternoon of postoperative day three
  The cumulative number of days (n) with a positive delirium screen will be calculated for all participants
Patient-Reported Quality of Recovery | Preoperative baseline through postoperative day three afternoon
  Assessed via the 15-item Quality of Recovery Score (n, 0-150, with higher number indicating better quality of recovery from the patient perspective)
Sedation | Preoperative baseline through postoperative day three afternoon
  Any positive screen based on the Richmond Agitation Sedation Scale (RASS; n, -5 to +4). Scores from -5 to -2 will count as a positive screen for sedation.
Agitation | Preoperative baseline through postoperative day three afternoon
  Any positive screen based on the Richmond Agitation Sedation Scale (RASS; n, -5 to +4). Scores from +2 to +4 will count as a positive screen for agitation
Headache | Preoperative baseline through postoperative day three afternoon
  Headache severity will be assessed via 10-centimeter visual analog scale (0-100 mm, with higher score indicating more severe headache)
Cumulative Opioid Consumption | Day of surgery through postoperative day three afternoon
  Postoperative opioid consumption, oral morphine equivalents (mg)

OTHER OUTCOMES:
Anesthetic Emergence | Duration of time from surgical dressing completion to anesthetic emergence (min); generally expected to be between 10 and 60 minutes
  Time (minutes) from surgical closure to extubation
Pulmonary Complications | From extubation until end of postanesthesia care unit stay
  Composite outcome (yes/no) of any of the following: airway adjunct use, unplanned continuous positive airway pressure device, unplanned humidified high-flow oxygen, need for bag-mask ventilation, or reintubation
Hospital Length of Stay | Morning of surgery until day of hospital discharge, up to 30 days
  Total number of days (n) spent in the hospital, up to 30 days
Discharge Disposition | Day of hospital discharge, up to 30 days
  Proportion of patients in each group (%) discharged somewhere other than home (e.g., Long-Term Care Facility), up to 30 days
30-Day Cognitive Function | 30 days after hospital discharge
  Cognitive function score based on the Montreal Cognitive Assessment (n, 0-30, with higher scores reflecting higher cognitive function)
30-Day Physical Function | 30 days after hospital discharge
  Physical function score based on the Patient Reported Outcomes Measurement Information System (PROMIS) Physical Function 10a score (n, 10-50, with higher score indicating better physical function)

CONTACTS AND LOCATIONS:
Overall Officials: Phillip Vlisides, MD, Principal Investigator — Assistant Professor of Anesthesiology
Locations (1):
- Michigan Medicine, Ann Arbor, Michigan, United States

IPD SHARING:
Plan to Share IPD: Yes
Clinical and electroencephalographic data will be preserved and made available for sharing. Data will be saved in various formats, such as comma-separated values (CSV), open document format (ODF), and European Data Format (EDF) for waveform data. Software programs designed to accommodate electroencephalographic waveform data (e.g., MATLAB) will be required for data access and analysis. Specific software and coding recommendations can be made available upon data sharing request.
  Any data not permitted to be shared, as specified in written informed consent documents, will be withheld. Likewise, no data will be shared that may compromise the safety or privacy of participants, and no data will be shared that would violate local, state, or federal laws or policies (including the Health Insurance Portability and Accountability Act). All data will be de-identified.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Scientific data will be made available after primary trial manuscripts (for both clinical and electroencephalographic data) are accepted for publication. Data will be made available for as long as possible in compliance with National Institutes of Health and University of Michigan policies.
Access Criteria: Data will be shared upon execution of Data Use Agreements in compliance with University of Michigan policies and procedures. Interested researchers will need to contact the study PI (Dr. Vlisides) for obtaining data via Data Use Agreement. All data will be shared upon reasonable request after primary trial manuscripts are published.

REFERENCES:
- [Background] Vlisides PE, Li D, McKinney A, Brooks J, Leis AM, Mentz G, Tsodikov A, Zierau M, Ragheb J, Clauw DJ, Avidan MS, Vanini G, Mashour GA. The Effects of Intraoperative Caffeine on Postoperative Opioid Consumption and Related Outcomes After Laparoscopic Surgery: A Randomized Controlled Trial. Anesth Analg. 2021 Jul 1;133(1):233-242. doi: 10.1213/ANE.0000000000005532. PMID 33939649
- [Background] Kim H, McKinney A, Brooks J, Mashour GA, Lee U, Vlisides PE. Delirium, Caffeine, and Perioperative Cortical Dynamics. Front Hum Neurosci. 2021 Dec 20;15:744054. doi: 10.3389/fnhum.2021.744054. eCollection 2021. PMID 34987367
- [Derived] Vlisides PE, Ragheb J, McKinney A, Mentz G, Runstadler N, Martinez S, Jewell E, Lee U, Vanini G, Schmitt EM, Inouye SK, Mashour GA. Caffeine, Postoperative Delirium And Change In Outcomes after Surgery (CAPACHINOS)-2: protocol for a randomised controlled trial. BMJ Open. 2023 May 15;13(5):e073945. doi: 10.1136/bmjopen-2023-073945. PMID 37188468